CLINICAL TRIAL: NCT05924802
Title: Physiological Effects of Dietary Supplement Ketone Ester on the Heart
Brief Title: Physiological Effects Ketone Ester in Heart
Acronym: KEHeart
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Christopher Nguyen, Director, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-570
Record Dates: First submitted 2023-06-09; First posted 2023-06-29 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: Placebo vs intervention group. Ketone ester is NOT a drug and only used to see the physiological effects on the heart.
Who Masked: Participant, Investigator
Masking Description: Both participant and investigators will be blinded. A representative in the center will be in charge of maintaining encrypted key.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo given that mimics taste, weight, and size of the interventional supplement mirroring the same time points as the ketone ester supplement group. Mirrored imaging with MRI as well.
  Interventions: Dietary Supplement: Placebo
- Ketone ester supplement (Experimental): Ketone ester given daily for 12 weeks and scanned before and after intervention with MRI.
  Interventions: Dietary Supplement: Ketone Ester

INTERVENTIONS:
Dietary Supplement: Ketone Ester — Added to water or lemonade 3 times per day.
  Other Names: delta G
  Arms: Ketone ester supplement
Dietary Supplement: Placebo — Added to water or lemonade 3 times per day.
  Arms: Placebo

SUMMARY:
The study is aimed to phenotype with cardiac MRI the physiological effects of ketone esters on the heart. Patients with heart failure will be recruited and given ketone esters or placebo in a randomized fashion. Cardiac MRI will be performed at baseline and after 12weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* heart failure EF < 40%

Exclusion Criteria:

* Claustrophobia
* Contraindicated implanted device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction | Pre-intervention and up to 12 weeks after intervention
  Measured with cardiac MRI the left ventricular ejection fraction at two points and then delta is calculated

SECONDARY OUTCOMES:
Change in Creatine concentration | Pre-intervention and up to 12 weeks after intervention
  Measured with cardiac MRI the creatine concentration at two points and then delta is calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Innovation Research Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yurista SR, Matsuura TR, Sillje HHW, Nijholt KT, McDaid KS, Shewale SV, Leone TC, Newman JC, Verdin E, van Veldhuisen DJ, de Boer RA, Kelly DP, Westenbrink BD. Ketone Ester Treatment Improves Cardiac Function and Reduces Pathologic Remodeling in Preclinical Models of Heart Failure. Circ Heart Fail. 2021 Jan;14(1):e007684. doi: 10.1161/CIRCHEARTFAILURE.120.007684. Epub 2020 Dec 28. PMID 33356362
- [Background] Yurista SR, Eder RA, Welsh A, Jiang W, Chen S, Foster AN, Mauskapf A, Tang WHW, Hucker WJ, Coll-Font J, Rosenzweig A, Nguyen CT. Ketone ester supplementation suppresses cardiac inflammation and improves cardiac energetics in a swine model of acute myocardial infarction. Metabolism. 2023 Aug;145:155608. doi: 10.1016/j.metabol.2023.155608. Epub 2023 Jun 1. PMID 37268056